CLINICAL TRIAL: NCT06291025
Title: Efficacy and Safety of Immunosuppression, Caplacizumab and Plasma Infusion Without Therapeutic Plasma Exchange in Immune-mediated Thrombotic Thrombocytopenic Purpura: Multicentric Non-inferiority Single-arm Study
Acronym: PEX-FREE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/0374/HP
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Thrombotic Microangiopathies
MeSH Terms: conditions — Thrombotic Microangiopathies

STUDY DESIGN:
Intervention Model Description: This trial is prospective, non-comparative, non-inferiority, single-arm, multicentric, national.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEX-FREE (Experimental): Replacing daily PEX with daily plasma infusions (ie. Quarantine fresh frozen plasma (PFC-Se), solvent detergent/viral inactivated plasma (PFC-SD = OCTAPLASLG) or amotosalen-inactivated plasma (PFC-IA); volume 15mL/kg/day).
  Interventions: Procedure: PEX-FREE

INTERVENTIONS:
Procedure: PEX-FREE — The study/experimental procedure consists in replacing daily PEX with daily plasma infusions (ie. Quarantine fresh frozen plasma (PFC-Se), solvent detergent/viral inactivated plasma (PFC-SD = OCTAPLASLG) or amotosalen-inactivated plasma (PFC-IA); volume 15mL/kg/day).
  Other Names: PEX-FREE procedure

SUMMARY:
Immune thrombotic thrombocytopenic purpura (iTTP) is caused by a severe, autoantibody-mediated deficiency of ADAMTS13 leading to an accumulation of ultra-large von Willebrand factor multimers in plasma and finally to microthrombi in blood vessels. The current standard of care of iTTP consists in the triple association of daily plasma exchange (PEX, 60 ml/kg/day), immunosuppressive agents and anti-adhesive treatment (Caplacizumab). Our group recently reported the outcome of 90 patients with iTTP treated with this triple association and when compared to historical patients, the triplet regimen prevented death, refractoriness and exacerbations. Likewise, plasma volumes were reduced by 2 to 3-fold and we could reduce the median number of PEX sessions from 13 to 6. PEX is an invasive and time-consuming procedure, associated with catheter and plasma-related complications ranging from 22% to 30%. Consequently, to alleviate the burden of care in iTTP, using a regimen without PEX would represent a major and topical goal. Attempts to treat patients with plasma infusion (PI) without PEX were previously reported and provided evidence that large volumes of PI (20-30 ml/kg/day) improved the initial outcome of iTTP. However, fluid overload occurred in most cases after 5-7 days, limiting the feasibility of this strategy. Nevertheless, the recent availability of caplacizumab opens the perspective of treating patients with plasma for a shorter period. Recently, strategies without PEX have been carried out in Jehovah's Witnesses with iTTP [5]. Impressively, improvement was rapid and comparable to those provided with a standard PEX-based treatment. Additionally, a treatment combining caplacizumab and immunosuppression only was successfully performed in six iTTP patients with severe neurologic and/or cardiac involvement. The rapid and durable improvement provides evidence that a regimen without plasma seems feasible. However, we consider that robust data are still lacking to completely remove plasmatherapy from iTTP management. Based on these statements, we wish here to address the efficacy and safety of a PEX-free regimen, combining PI only (15 ml/kg/day), corticosteroids/rituximab, and caplacizumab.

DETAILED DESCRIPTION:
Immune thrombotic thrombocytopenic purpura (iTTP) is caused by a severe, autoantibody-mediated deficiency of ADAMTS13 leading to an accumulation of ultra-large von Willebrand factor multimers in plasma and finally to microthrombi in blood vessels. The current standard of care of iTTP consists in the triple association of daily plasma exchange (PEX, 60 ml/kg/day), immunosuppressive agents and anti-adhesive treatment (Caplacizumab). Our group recently reported the outcome of 90 patients with iTTP treated with this triple association and when compared to historical patients, the triplet regimen prevented death, refractoriness and exacerbations. Likewise, plasma volumes were reduced by 2 to 3-fold and we could reduce the median number of PEX sessions from 13 to 6. PEX is an invasive and time-consuming procedure, associated with catheter and plasma-related complications ranging from 22% to 30%. Consequently, to alleviate the burden of care in iTTP, using a regimen without PEX would represent a major and topical goal. Attempts to treat patients with plasma infusion (PI) without PEX were previously reported and provided evidence that large volumes of PI (20-30 ml/kg/day) improved the initial outcome of iTTP. However, fluid overload occurred in most cases after 5-7 days, limiting the feasibility of this strategy. Nevertheless, the recent availability of caplacizumab opens the perspective of treating patients with plasma for a shorter period. Recently, strategies without PEX have been carried out in Jehovah's Witnesses with iTTP [5]. Impressively, improvement was rapid and comparable to those provided with a standard PEX-based treatment. Additionally, a treatment combining caplacizumab and immunosuppression only was successfully performed in six iTTP patients with severe neurologic and/or cardiac involvement. The rapid and durable improvement provides evidence that a regimen without plasma seems feasible. However, we consider that robust data are still lacking to completely remove plasmatherapy from iTTP management. Based on these statements, we wish here to address the efficacy and safety of a PEX-free regimen, combining PI only (15 ml/kg/day), corticosteroids/rituximab, and caplacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years;
* Clinical diagnosis of iTTP based on standard clinical and laboratory criteria (French Score ≥ 2): i.e., thrombotic microangiopathy syndrome with platelet count ≤ 30 G/L and serum creatinine ≤ 200 μmol/L; it is not necessary to have the laboratory result confirming the severe ADAMTS13 deficiency for inclusion of patient [32] (For patient with previous TTPflare, French score can be < 2);
* Patient having read and understood the information letter and signed the Informed Consent Form. If the patient is unable to express his consent, the consent will be signed by his representative ((1) the trusted person, or failing that, (2) a family member, or (3) a close relative of the person concerned). In this case, consent to continue the study will subsequently be requested from the patient (article L1122-1-1 of the CSP);
* Patient affiliated with, or beneficiary of a social security (national health insurance) plan;
* For women:

  * Women of childbearing potential :

    * Effective contraception according to WHO definition (estrogen-progestin or intrauterine device or tubal ligation) since at least 1 month and;
    * Negative blood pregnancy test;
  * Women surgically sterile (absence of ovaries and/or uterus);
  * Postmenopausal women (non-medically induced amenorrhea for at least 12 months prior to the inclusion visit).

Exclusion Criteria:

* Platelet count > 100 G/L before plasma treatment;
* Patients with a French score < 2 (a serum creatinine level > 200 μmol/L and/or with a platelet count > 30 G/L), in order to exclude possible cases of hemolytic uremic syndrome (except for patient with previous TTPflare, French score can be < 2);
* Other known causes of cytopenias and/or organ failure including but not limited to: uncontrolled cancer, chemotherapy, transplant, drugs, HIV at AIDS stage;
* Patients with a severe neurological disorder i.e. seizure, coma, focal deficiency, trouble of consciousness;
* Pregnant women (positive result from a blood pregnancy test) or patients with an imminent project of pregnancy; breastfeeding women (due to lack of pharmacological data for caplacizumab during pregnancy and breastfeeding);
* Weight > 100KG;
* Congenital TTP;
* Clinically significant active bleeding or high risk of bleeding (excluding thrombocytopenia);
* Chronic treatment with anticoagulant that cannot be interrupted safely, including but not limited to: vitamin K antagonists, direct oral anticoagulant, low molecular weight heparin or heparin;
* Malignant hypertension;
* Contra-indication to CABLIVI 10 mg powder and solvent for solution for injection: hypersensitivity to caplacizumab or to any of the excipients;
* Contra-indication to Plasma treatment;
* Contra-indication to corticosteroid (= ((methyl)prednisone or (methyl)prednisolone)) or excipients;
* Contra-indication to rituximab or excipients and to its premedication;
* Person deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision);
* Participation in another drug interventional clinical trial within 30 days prior to inclusion and during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of a PEX-FREE regimen in adults with iTTP as assessed by the proportion of participants day-30 post-plasma therapy death, refractoriness, exacerbation or an ADAMTS13 activity < 20%. | 30 days
  Complete plasma infusion treatment and clinical remission at day 30 defined by both lack of occurrence of any of the four events during the 30 days post plasma infusion procedure

IPD SHARING:
Plan to Share IPD: No